CLINICAL TRIAL: NCT06463184
Title: A Phase 1, Open-Label Window-of-Opportunity Study to Assess the Pharmacokinetics, Pharmacodynamics and Central Nervous System (CNS) Penetration of Xevinapant in Preoperative Subjects With Recurrent High-Grade Glioma (rHGG)
Brief Title: Study to Assess Xevinapant in Preoperative Subjects With Recurrent High-Grade Glioma (rHGG)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: funding issues
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22511
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Recurrent High-grade Glioma
MeSH Terms: conditions — Glioma | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xevinapant Treatment (Experimental): Participants will be given a course of orally administered Xevinapant at 400 mg once daily for 4 consecutive days, prior to undergoing clinically indicated tumor resection.
  Interventions: Drug: Xevinapant

INTERVENTIONS:
Drug: Xevinapant — Xevinapant is an investigational medication, taken orally, that promotes cancer cell death via apoptosis.
  Other Names: Debio 1143

SUMMARY:
Researchers will investigate the ability of Xevinapant to cross the blood-brain barrier and exert anti-tumor effects on rHGG through activation of apoptosis. Researchers hypothesize that oral administration of Xevinapant has acceptable safety and tolerability in patients with recurrent HGG and demonstrate pharmacokinetic and pharmacodynamic effects in HGG tumors. To that end, Researchers will engage in a phase I "window of opportunity" translational clinical trial in patients undergoing a clinically-indicated craniotomy for resection of recurrent tumors to evaluate the impact of treatment on rHGG.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age (or based on the country legal age limit for adults) on day of signing the Informed Consent Form (ICF).
* Patient must have histologically confirmed diagnosis of: WHO grade III or IV glioma or glioblastoma or gliosarcoma. This definition also includes anaplastic astrocytoma, anaplastic oligodendroglioma, and anaplastic mixed glioma.
* Radiographic evidence of tumor recurrence.
* Contrast enhancing tumor that is amenable to surgical resection
* Patient must be able to understand and willing to sign an informed consent.
* Patient must have Karnofsky performance status (KPS) of ≥70 or Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
* Able to swallow liquids or has an adequately functioning feeding tube, gastrostomy or jejunostomy placed.
* Adequate hematologic, renal, and hepatic function as indicated by the protocol.
* Women of childbearing potential (according to recommendations of the Clinical Trial Facilitation Group) must have a negative serum pregnancy test at screening and must not be breastfeeding. Women of childbearing potential must agree to use highly effective contraceptive method(s) from ICF signature to 6 months after the last administration of chemotherapy or 3 months after last dose of xevinapant. Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use condom and spermicide from ICF signature to 6 months after the last administration of chemotherapy or 3 months after the last dose of xevinapant. Because male condom and spermicide is not a highly effective contraception method, it is required that female partners of a male study subject use highly effective contraceptive method(s) throughout this period. Male subjects must refrain from donating sperm during the clinical study and for 6 months after the last administration of chemotherapy or 3 months after the last dose of xevinapant. If not done previously, cryopreservation of sperm prior to receiving chemotherapy or xevinapant is advised to male patients with a desire to have children.
* Subject may or may not have archived primary tumor biopsies or surgical specimens, or biopsies of recurrence tumor for exploratory translational studies. We will enroll at least 4-6 subjects with archival tissue for biomarker/PD studies. For those with archival tissue, at least 10 unstained FFPE tissue slides or a tissue block should be available for enrollment. If less material is available, subject could still be eligible after discussion with the Principal Investigator who will assess and confirm that there is sufficient material for key evaluations.

Exclusion Criteria:

* Use within 14 days prior to randomization or requirement for ongoing treatment with any drug(s) on the prohibited medication list (see "prohibited concomitant drugs" in section 6.5).
* Known history of infection with HIV. If unknown history of HIV, an HIV screening test is to be performed and subjects with positive serology for HIV-1/2 must be excluded.
* Known chronically active HBV or HCV infection. If unknown status, the following tests are to be performed and subjects with positive serology must be excluded: A) HBV screening tests: both HBV sAg and Anti-HepB core IgG. B) HCV screening tests: both HCV-antibody and positive viral load HCV-RNA by PCR.
* Other infections (viral and/or bacterial and/or mycotic) requiring systemic treatment.
* Live-attenuated vaccinations within 30 days prior to first investigational treatment administration.
* Ongoing uncontrolled infection requiring intravenous antibiotic therapy within 1 week prior to randomization.
* Documented weight loss of >10% during the last 4 weeks prior to randomization (unless adequate measures are undertaken for nutritional support), OR plasmatic albumin < 3.0 g/dL. No albumin transfusions are allowed within 2 weeks before randomization.
* Active uncontrolled inflammatory disease (including rheumatoid arthritis, systemic lupus erythematosus, Sjögren syndrome, severe extensive psoriasis, and other autoimmune diseases) requiring ongoing treatment with anti-TNF medication.
* Any concomitant medication known to prolong the QT interval that cannot be discontinued or replaced by safe alternative medication within 7 days prior to start of treatment.
* Known allergy to Xevinapant or any excipient known to be present in active formulation.
* Non-compensated or symptomatic liver cirrhosis (Child-Pugh score: B or C).
* Treatment with an investigational agent or use of an investigational device within 4 weeks of the first dose of study treatment.
* Known gastrointestinal disorder with clinically established malabsorption syndrome and major gastrointestinal surgery that may limit oral absorption.
* Active gastrointestinal bleeding, or any other uncontrolled bleeding requiring more than 2 red blood cell transfusions or 4 units of packed red blood cells within 4 weeks prior to randomization.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following: A) Ongoing or history of uncontrolled or symptomatic ischemic myocardiopathy within 6 months prior to randomization. B) Known left ventricular ejection fraction <50%, left ventricular hypertrophy, ventricular arrhythmias, bradycardia (heart rate < 50 bpm). C) History of myocardial infarction, or severe/unstable angina, within 6 months prior to randomization. D) New York Heart Association grade ≥ 3 congestive heart failure. E) Congenital long QT syndrome. F) Family history of long QT syndrome. G) Symptomatic pulmonary embolism within 6 months prior to randomization. H) Ongoing or known history of transient ischemic attacks or stroke within 6 months prior to randomization. I) QTc using Fridericia's formula (QTcF) interval > 470 ms.
* Symptomatic pulmonary disease requiring continuous or intermittent oxygen supply.
* History of another malignancy within the last 3 years prior to randomization, with the exception of completely resected non-melanoma cell skin cancer outside the head and neck area or completely resected stage I breast cancer, or completely resected in-situ non-muscular invasive bladder, cervix and/or uterine carcinomas.
* Any ongoing condition or disorder, before randomization, including drug(s) or alcohol abuse, which in the judgment of the Investigator would make the patient inappropriate for entry into the study or precluding his/her ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of Xevinapant | Within 48 hours of last dose of Xevinapant.
  Concentration of unbound Xevinapant in brain tumor tissue in an exploratory manner (within contrast enhancing tumor as well as non-enhancing tumor, wherever possible) at the time of planned salvage resection.
Concentration max (Cmax) | Within 48 hours of last dose of Xevinapant.
  Maximum observed plasma concentration of Xevinapant.

SECONDARY OUTCOMES:
Occurrence of AE's and SAE's | Up to 12 months.
  The number of patients who experience AE's and SAE's.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Etame, MD, PhD, Principal Investigator — Moffitt Cancer Center